CLINICAL TRIAL: NCT00678639
Title: Randomized Cost Comparison of Cardiac MRI Use in ED Patients With Chest Pain
Brief Title: Cost Comparison of Cardiac Magnetic Resonance Imaging (MRI) Use in Emergency Department (ED) Patients With Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00004120
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Results first posted 2010-04-28 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: ACS; Acute Coronary Syndrome; Chest pain; Cardiac MRI; CMR; Risk Stratification; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies | interventions — Family Characteristics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Emergency Department (ED) Observation unit (Experimental): Emergency Department observation unit- Cardiac Magnetic Resonance Imaging (MRI) Protocol. Patients will be transferred to the observation unit and undergo a stress cardiac MRI evaluation.
  Interventions: Other: Observation unit care, coupled with cardiac MRI
- Usual care (No Intervention): This is the comparison arm. Patients are admitted to the hospital and undergo usual care.

INTERVENTIONS:
Other: Observation unit care, coupled with cardiac MRI — After Emergency Department (ED) evaluation, patients are randomized to Observation unit care or standard inpatient care. Patients in the observation unit will also undergo a stress cardiac MRI. Patients in the usual care arm may undergo any desired testing, including cardiac MRI, as determined by their treating physician.
  Arms: Emergency Department (ED) Observation unit

SUMMARY:
The purpose of this study is to investigate the best way to evaluate patients with chest pain in the emergency department. It compares receiving treatment in an observation unit with admission to the hospital. Patients treated in the observation unit will undergo cardiac Magnetic Resonance Imaging (MRI) testing. Patients treated with hospital admission will undergo the testing their doctor determines is best for them. All patients will undergo follow up to find out if they have had any heart related events.

DETAILED DESCRIPTION:
Almost half of patients presenting to the Emergency Department (ED) with possible cardiac chest pain are at intermediate risk for short term death or infarction. Most are admitted to the hospital for serial ECG's, cardiac biomarkers, cardiology consultation, and stress testing or coronary angiogram. However, the 2007 ACC/AHA guidelines suggest that these patients can be managed in an observation unit (OU). Recently, cardiac magnetic resonance imaging (CMR) has proven more accurate than traditional testing modalities for the diagnosis of acute coronary syndrome (ACS), and has also received endorsement from the American College of Cardiology (ACC)/American Heart Association (AHA) guidelines. Immediate application of CMR in an OU may improve health care utilization compared to standard hospital admission for intermediate risk patients.

Research hypotheses:

1. Patients in an OU CMR protocol will have lower cost for the index hospitalization than standard care.
2. An OU CMR protocol for patients with intermediate risk chest pain will significantly improve the frequency of correct cardiovascular admission decisions when compared to standard care.

Methods summary:

110 ED patients at intermediate risk for short-term death or infarction, with nondiagnostic Electrocardiograms (ECG) and normal initial cardiac biomarkers, will be randomized to standard care or OU CMR protocols. Subjects in the OU CMR protocol will undergo CMR perfusion and stress testing, followed by serial biomarkers. Standard care subjects will be admitted for usual cardiac testing. ACS (infarction, death, coronary revascularization, unstable angina) will be assessed by evaluation of hospital course and phone follow-up at 30 days. Cost of hospital care will be compared among groups.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age at the time of enrollment
* Chest discomfort or other symptoms consistent with possible Acute Coronary Syndrome (ACS) as indicated by the treating physician after obtaining an Electrocardiogram (ECG) and cardiac biomarkers for the patient's evaluation
* Patient requires an inpatient evaluation for their chest pain
* The treating physician feels the patient could be discharged home if cardiac disease was excluded
* Thrombolysis in Myocardial Infarction (TIMI) risk score ≥ 2 OR physician clinical impression of intermediate or high likelihood that the symptoms represent ACS
* Negative pregnancy test (if sexually active, female, and of childbearing age)

Exclusion Criteria:

* Initial troponin I > 1.0 ng/ml
* New ST-segment elevation on any electrocardiogram (≥ 1 mV)
* New ST-segment depression on any electrocardiogram (≥ 2 mV)
* Unable to lie flat
* Hypotension (systolic < 90 mm Hg)
* Contra-indications to MRI(Pacemaker, defibrillator, cerebral aneurysm clips, metallic ocular foreign body, implanted devices, claustrophobia)
* Patient refusal of medical record review and telephone follow-up at 30 days
* Terminal diagnosis with life expectancy less than 3 months
* Pregnancy per patient report or positive pregnancy test (Center for Medicare & Medicaid Services (CMS) exclusion criteria)
* Renal insufficiency(done prior to enrollment)or end stage renal disease
* Chronic liver disease (ex. hepatitis, cirrhosis)
* History of liver, heart, or kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick D Miller, MD, Principal Investigator — WFUBMC
Locations (1):
- Wake Forest University Baptist Medical Center - Emergency Department, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Gomberg-Maitland M, Murphy SA, Moliterno DJ, Cannon CP. Are we appropriately triaging patients with unstable angina? Am Heart J. 2005 Apr;149(4):613-8. doi: 10.1016/j.ahj.2004.09.035. PMID 15990742
- [Background] Desai AS, Solomon DH, Stone PH, Avorn J. Economic consequences of routine coronary angiography in low- and intermediate-risk patients with unstable angina pectoris. Am J Cardiol. 2003 Aug 15;92(4):363-7. doi: 10.1016/s0002-9149(03)00650-7. PMID 12914862
- [Background] Tatum JL, Jesse RL, Kontos MC, Nicholson CS, Schmidt KL, Roberts CS, Ornato JP. Comprehensive strategy for the evaluation and triage of the chest pain patient. Ann Emerg Med. 1997 Jan;29(1):116-25. doi: 10.1016/s0196-0644(97)70317-2. PMID 8998090
- [Background] Stowers SA, Eisenstein EL, Th Wackers FJ, Berman DS, Blackshear JL, Jones AD Jr, Szymanski TJ Jr, Lam LC, Simons TA, Natale D, Paige KA, Wagner GS. An economic analysis of an aggressive diagnostic strategy with single photon emission computed tomography myocardial perfusion imaging and early exercise stress testing in emergency department patients who present with chest pain but nondiagnostic electrocardiograms: results from a randomized trial. Ann Emerg Med. 2000 Jan;35(1):17-25. doi: 10.1016/S0196-0644(00)70100-4. PMID 10613936
- [Background] Calvin JE, Klein LW, VandenBerg EJ, Meyer P, Parrillo JE. Validated risk stratification model accurately predicts low risk in patients with unstable angina. J Am Coll Cardiol. 2000 Nov 15;36(6):1803-8. doi: 10.1016/s0735-1097(00)00977-3. PMID 11092647
- [Background] Robinson DJ, Woods PG, Snedeker CA, Lynch JH, Chambers K. A comparison trial for stratifying intermediate-risk chest pain: benefits of emergency department observation centers. Prev Cardiol. 2002 Winter;5(1):23-30. doi: 10.1111/j.1520-037x.2002.00550.x. PMID 11872988
- [Background] Committee on the Future of Emergency Care in the United States Health System. 2006. Hospital-Based Emergency Care: At the Breaking Point. Washington, DC: The National Academies Press.
- [Background] Ramakrishna G, Milavetz JJ, Zinsmeister AR, Farkouh ME, Evans RW, Allison TG, Smars PA, Gibbons RJ. Effect of exercise treadmill testing and stress imaging on the triage of patients with chest pain: CHEER substudy. Mayo Clin Proc. 2005 Mar;80(3):322-9. doi: 10.4065/80.3.322. PMID 15757012
- [Background] Conti A, Pieralli F, Sammicheli L, Camaiti A, Vanni S, Grifoni S, Dovellini E, Antoniucci D, Squillantini G, Mazzuoli F, Colombo G. Updated management of non-st-segment elevation acute coronary syndromes: selection of patients for low-cost care: an analysis of outcome and cost effectiveness. Med Sci Monit. 2005 Mar;11(3):CR100-8. PMID 15735561
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Committee to Update the 1997 Exercise Testing Guidelines. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). J Am Coll Cardiol. 2002 Oct 16;40(8):1531-40. doi: 10.1016/s0735-1097(02)02164-2. No abstract available. PMID 12392846
- [Background] Detrano R, Gianrossi R, Froelicher V. The diagnostic accuracy of the exercise electrocardiogram: a meta-analysis of 22 years of research. Prog Cardiovasc Dis. 1989 Nov-Dec;32(3):173-206. doi: 10.1016/0033-0620(89)90025-x. No abstract available. PMID 2530605
- [Background] Gianrossi R, Detrano R, Mulvihill D, Lehmann K, Dubach P, Colombo A, McArthur D, Froelicher V. Exercise-induced ST depression in the diagnosis of coronary artery disease. A meta-analysis. Circulation. 1989 Jul;80(1):87-98. doi: 10.1161/01.cir.80.1.87. PMID 2661056
- [Background] Geleijnse ML, Fioretti PM, Roelandt JR. Methodology, feasibility, safety and diagnostic accuracy of dobutamine stress echocardiography. J Am Coll Cardiol. 1997 Sep;30(3):595-606. doi: 10.1016/s0735-1097(97)00206-4. PMID 9283514
- [Background] Klocke FJ, Baird MG, Lorell BH, Bateman TM, Messer JV, Berman DS, O'Gara PT, Carabello BA, Russell RO Jr, Cerqueira MD, St John Sutton MG, DeMaria AN, Udelson JE, Kennedy JW, Verani MS, Williams KA, Antman EM, Smith SC Jr, Alpert JS, Gregoratos G, Anderson JL, Hiratzka LF, Faxon DP, Hunt SA, Fuster V, Jacobs AK, Gibbons RJ, Russell RO; American College of Cardiology; American Heart Association; American Society for Nuclear Cardiology. ACC/AHA/ASNC guidelines for the clinical use of cardiac radionuclide imaging--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (ACC/AHA/ASNC Committee to Revise the 1995 Guidelines for the Clinical Use of Cardiac Radionuclide Imaging). J Am Coll Cardiol. 2003 Oct 1;42(7):1318-33. doi: 10.1016/j.jacc.2003.08.011. No abstract available. PMID 14522503
- [Background] Hilton TC, Thompson RC, Williams HJ, Saylors R, Fulmer H, Stowers SA. Technetium-99m sestamibi myocardial perfusion imaging in the emergency room evaluation of chest pain. J Am Coll Cardiol. 1994 Apr;23(5):1016-22. doi: 10.1016/0735-1097(94)90584-3. PMID 8144763
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Udelson JE, Beshansky JR, Ballin DS, Feldman JA, Griffith JL, Handler J, Heller GV, Hendel RC, Pope JH, Ruthazer R, Spiegler EJ, Woolard RH, Selker HP. Myocardial perfusion imaging for evaluation and triage of patients with suspected acute cardiac ischemia: a randomized controlled trial. JAMA. 2002 Dec 4;288(21):2693-700. doi: 10.1001/jama.288.21.2693. PMID 12460092
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Bashore TM, Bates ER, Berger PB, Clark DA, Cusma JT, Dehmer GJ, Kern MJ, Laskey WK, O'Laughlin MP, Oesterle S, Popma JJ, O'Rourke RA, Abrams J, Bates ER, Brodie BR, Douglas PS, Gregoratos G, Hlatky MA, Hochman JS, Kaul S, Tracy CM, Waters DD, Winters WL Jr; American College of Cardiology. Task Force on Clinical Expert Consensus Documents. American College of Cardiology/Society for Cardiac Angiography and Interventions Clinical Expert Consensus Document on cardiac catheterization laboratory standards. A report of the American College of Cardiology Task Force on Clinical Expert Consensus Documents. J Am Coll Cardiol. 2001 Jun 15;37(8):2170-214. doi: 10.1016/s0735-1097(01)01346-8. No abstract available. PMID 11419904
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Karha J, Gibson CM, Murphy SA, Dibattiste PM, Cannon CP; TIMI Study Group. Safety of stress testing during the evolution of unstable angina pectoris or non-ST-elevation myocardial infarction. Am J Cardiol. 2004 Dec 15;94(12):1537-9. doi: 10.1016/j.amjcard.2004.08.033. PMID 15589011
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Moher D, Rennie D, de Vet HC, Lijmer JG; Standards for Reporting of Diagnostic Accuracy. The STARD statement for reporting studies of diagnostic accuracy: explanation and elaboration. Ann Intern Med. 2003 Jan 7;138(1):W1-12. doi: 10.7326/0003-4819-138-1-200301070-00012-w1. PMID 12513067
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Antman EM, Cohen M, Bernink PJ, McCabe CH, Horacek T, Papuchis G, Mautner B, Corbalan R, Radley D, Braunwald E. The TIMI risk score for unstable angina/non-ST elevation MI: A method for prognostication and therapeutic decision making. JAMA. 2000 Aug 16;284(7):835-42. doi: 10.1001/jama.284.7.835. PMID 10938172
- [Background] Hundley WG, Hamilton CA, Thomas MS, Herrington DM, Salido TB, Kitzman DW, Little WC, Link KM. Utility of fast cine magnetic resonance imaging and display for the detection of myocardial ischemia in patients not well suited for second harmonic stress echocardiography. Circulation. 1999 Oct 19;100(16):1697-702. doi: 10.1161/01.cir.100.16.1697. PMID 10525488
- [Background] Hundley WG, Morgan TM, Neagle CM, Hamilton CA, Rerkpattanapipat P, Link KM. Magnetic resonance imaging determination of cardiac prognosis. Circulation. 2002 Oct 29;106(18):2328-33. doi: 10.1161/01.cir.0000036017.46437.02. PMID 12403662
- [Background] Hundley WG, Hamilton CA, Rerkpattanapipat P. Magnetic resonance imaging assessment of cardiac function. Curr Cardiol Rep. 2003 Jan;5(1):69-74. doi: 10.1007/s11886-003-0040-1. PMID 12493163
- [Background] Puskas JD, Williams WH, Mahoney EM, Huber PR, Block PC, Duke PG, Staples JR, Glas KE, Marshall JJ, Leimbach ME, McCall SA, Petersen RJ, Bailey DE, Weintraub WS, Guyton RA. Off-pump vs conventional coronary artery bypass grafting: early and 1-year graft patency, cost, and quality-of-life outcomes: a randomized trial. JAMA. 2004 Apr 21;291(15):1841-9. doi: 10.1001/jama.291.15.1841. PMID 15100202
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764
- [Background] Goodacre S, Nicholl J, Dixon S, Cross E, Angelini K, Arnold J, Revill S, Locker T, Capewell SJ, Quinney D, Campbell S, Morris F. Randomised controlled trial and economic evaluation of a chest pain observation unit compared with routine care. BMJ. 2004 Jan 31;328(7434):254. doi: 10.1136/bmj.37956.664236.EE. Epub 2004 Jan 14. PMID 14724129
- [Background] Miller CD, Lindsell CJ, Fermann GJ, et al. After the First Negative Troponin: Distinguishing Patients with Evolving Myocardial Infarctions from Those Without Infarction in Emergency Department Patients with Chest Pain. Annals of Emergency Medicine 2005;46(3, Supplement 1):114-5.
- [Background] Geleijnse ML, Elhendy A, Kasprzak JD, Rambaldi R, van Domburg RT, Cornel JH, Klootwijk AP, Fioretti PM, Roelandt JR, Simoons ML. Safety and prognostic value of early dobutamine-atropine stress echocardiography in patients with spontaneous chest pain and a non-diagnostic electrocardiogram. Eur Heart J. 2000 Mar;21(5):397-406. doi: 10.1053/euhj.1999.1860. PMID 10666354
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Derived] Miller CD, Hwang W, Case D, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Hundley WG. Stress CMR imaging observation unit in the emergency department reduces 1-year medical care costs in patients with acute chest pain: a randomized study for comparison with inpatient care. JACC Cardiovasc Imaging. 2011 Aug;4(8):862-70. doi: 10.1016/j.jcmg.2011.04.016. PMID 21835378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the emergency department January 2008 - March 2009.
Pre-assignment Details: Once consented, no participants were excluded from the trial prior to group assignment.
Groups:
- Emergency Department (ED) Observation Unit: Emergency Department observation unit - Cardiac Magnetic Resonance Imaging (MRI) Protocol. Patients will be transferred to the observation unit and undergo a stress cardiac MRI evaluation.
Period: Overall Study
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Started | 53 | 57
Hospital Discharge | 53 | 57
Completed | 51 | 57
Not Completed | 2 | 0
Not completed — Lost to Follow-up at 30 days | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care | Total
Number analyzed (Participants) | 53 | 57 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 92
  >=65 years | 8 | 10 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 25 | 30 | 55
Region of Enrollment [Number; unit: participants]
  United States | 53 | 57 | 110

OUTCOME MEASURES:

1. Primary Outcome: Cost of Index Hospitalization
Description: Index hospitalization refers to the hospital visit during which the participant was enrolled in the trial. The primary outcome is examining the cost for this visit.
Time Frame: Emergency Department (ED) arrival through hospital discharge, median length of stay was 28.1 hours
Population: All participants were analyzed based on intention to treat.
Measure: Median (Inter-Quartile Range); unit: US Dollars
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Number analyzed (Participants) | 53 | 57
US Dollars | 2062 [1918 to 2367] | 2680 [2408 to 3448]
Statistical Analysis 1: Comparison: Emergency Department (ED) Observation Unit vs Usual Care; H0: The median costs are not different among the study groups. HA: The median cost is different among groups. Power calculation was based on detecting a mean cost difference of $2000. Data was found to be non-normally distributed and therefore nonparametric comparisons were implemented; Test type: Superiority or Other; Hodges-Lehmann (median cost difference); Distribution-free 95% CIs calculated using the method of Moses; Median cost difference = 588, 95% CI 2-sided [336 to 811] — Results favored a reduced cost in the OU-CMR group

2. Secondary Outcome: Correct Admission Decision, Based Upon the Reference Standard of Acute Coronary Syndrome (ACS) at 30 Days
Description: Participants with ACS and admitted or not experiencing ACS and discharged will be considered a correct admission decision. Remaining participants will be considered to have incorrect admission decisions.
Time Frame: 30 Days
Population: 4 participants (3 in the usual care group and 1 in the ED obs unit group) left Against Medical Advice (AMA) prior to completion of their evaluation and were excluded from this analysis. Analysis was per intention to treat.
Measure: Number; unit: Participants
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Number analyzed (Participants) | 52 | 54
Participants | 43 | 6
Statistical Analysis 1: Comparison: Emergency Department (ED) Observation Unit vs Usual Care; H0: There is no difference in correct cardiovascular admission decisions among groups. Ha: A difference exists among study groups. Sample size was based upon 47 analyzable participants per study arm were required to provide 88% power to detect a 30% difference in the outcome; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: The Number of Participants Randomized to the OU and Were Able to Complete CMR Imaging
Description: The number of participants able to complete the planned imaging sequences will be measured.
Time Frame: Emergency Department (ED) arrival through hospital discharge
Population: All participants randomized to the Observation Unit - Cardiac Magnetic Resonance Imaging (OU-CMR) arm were analyzed based on intention to treat.
Measure: Number; unit: Participants
Groups:
- Emergency Department (ED) Observation Unit: Emergency Department observation unit- Cardiac MRI Protocol. Patients will be transferred to the observation unit and undergo a stress cardiac MRI evaluation.
Arm/Group | Emergency Department (ED) Observation Unit
Number analyzed (Participants) | 53
Participants | 46

4. Secondary Outcome: Number of Participants Who Utilized the Indicated Health Care Procedures
Description: Measured as self report, assessed during telephone follow-up.
Time Frame: 30d, 3mo, 6mo, and 1 year
Population: Data reported through 30 days. Follow-up with participants is ongoing. Results will be updated once follow-up is complete.
Measure: Number; unit: Participants
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Number analyzed (Participants) | 53 | 57
Participants
  Cardiac related office visit | 7 | 4
  Cardiac related ED visit | 0 | 4
  Cardiac related hospitalization | 0 | 3
  Cardiac related procedures | 0 | 4
  Cardiac Catheterization | 0 | 3
  Stress Test | 0 | 1
  Resting Echocardiogram | 0 | 1

5. Secondary Outcome: Adverse Events During Magnetic Resonance Imaging (MRI) Scanning
Description: Any event leading to early termination of the MRI acquisition, or requiring intervention by a physician, will be considered an adverse event related to MRI, excluding physician termination of image acquisition due to concerns of cardiac ischemia.
Time Frame: Occuring in the MRI scanning suite or within 30 minutes of the last image acquisition.
Population: Only participants undergoing Cardiac MRI scanning are eligible for this endpoint. Only 49 of the 53 participants randomized to observation unit arm underwent CMR testing. Nine participants in the usual care arm underwent CMR testing.
Measure: Number; unit: Participants
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Number analyzed (Participants) | 49 | 9
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: The reported adverse event data was collected from participant enrollment through 90 days.
Description: Adverse event assessment is ongoing and will be updated when follow-up is complete.
Arm/Group | Emergency Department (ED) Observation Unit | Usual Care
Serious Adverse Events (participants affected / at risk) | 2/53 | 7/57
Other Adverse Events (participants affected / at risk) | 6/53 | 4/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emergency Department (ED) Observation Unit (N=53) | Usual Care (N=57)
Hospitalization for abdominal pain due to cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hospitalization for cerebral infarct (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization for chest pain (Cardiac disorders) | 0 (0) | 5 (6)
Hospitalization for chest pain and suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalization for neck surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emergency Department (ED) Observation Unit (N=53) | Usual Care (N=57)
Excessive cost of cardiac testing without Acute Coronary Syndrome (ACS) (Investigations) | 5 (5) | 1 (1)
Participant left before evaluation was completed (Social circumstances) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes